CLINICAL TRIAL: NCT06408272
Title: Electrical Impedance Tomography (EIT) for the Setting of High-pressure in Patients With Acute Respiratory Distress Syndrome (ARDS) on Time Controlled Adaptive Ventilation (TCAV).
Brief Title: Eit in ArdS for Tcav Setting (EAST Study)
Acronym: EAST
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI097
Record Dates: First submitted 2022-09-09; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: ARDS
Keywords: ARDS; TCAV; EIT; APRV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TCAV EIT: Patients with early ARDS, < 72h of Mechanical ventilation, under TCAV since one hour with EIT.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe form of acute respiratory failure. The therapeutic management is currently based on the treatment of the cause of ARDS, and on mechanical ventilation with positive expiratory pressure (PEEP). Another strategy that could be used is Time Controlled Adaptive Ventilation (TCAV) method based on ventilation using the airway pressure release ventilation (APRV) mode.

Electrical impedance tomography (EIT) allows individual, non-invasive, real-time, bedside, radiation-free imaging of an anteroposterior section of the right and left lungs, with global and regional dynamic analyses.

The aim of the study is to evaluate EIT for PHigh titration of TCAV.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a severe form of acute respiratory failure with a mortality rate of up to 35% for the most severe forms. The therapeutic management is currently based on the treatment of the cause of ARDS, and on mechanical ventilation with positive expiratory pressure (PEEP). Another strategy that could be used is Time Controlled Adaptive Ventilation (TCAV) method based on ventilation using the airway pressure release ventilation (APRV) mode.

The TCAV method is based on a prolonged THigh set at a constant pressure, creating a continuous positive pressure phase associated with a brief release during a TLow allowing the elimination of carbon dioxide and the creation of an intrinsic PEEP. With long high pressure phase this method could result in better recruitment but could also expose the patient to overdistention. While the TLow setting is well defined, level of PHigh is not standardized.

Electrical impedance tomography (EIT) allows individual, non-invasive, real-time, bedside, radiation-free imaging of an anteroposterior section of the right and left lungs, with global and regional dynamic analyses. Results of recent studies have highlighted the benefits of EIT, especially for ARDS patients in titrating PEEP in volume-controlled ventilation.

To date, no published study has evaluated EIT for PHigh titration using the TCAV method in patients with severe ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS patients with more than 24 hours of mechanical ventilation
* Under sedation with a Richmond Rating Scale less than or equal to -2.

Exclusion Criteria:

* Patients with a pacemaker or automatic implantable defibrillator
* Pregnant women.
* Contraindications to chest belt placement (e.g., spinal or thoracic recent surgery)
* Undrained pneumothorax, broncho-pleural fistula
* Hemodynamic instability (i.e., use of vasopressors at > 2 ug.kg.min of norepinephrine)
* Patients on mechanical ventilation during more than 7 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early moderate to severe ARDS under mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of collapsed units on EIT | through study completion an average of 1 day
  Percentage of collapsed lung areas measured at increasing levels of Phigh

SECONDARY OUTCOMES:
Percentage of overdistanded units | through study completion an average of 1 day
  Percentage of overdistanded units measured at increasing levels of Phigh

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu KOSZUTSKI, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided